CLINICAL TRIAL: NCT02946138
Title: A Prospective Phase II Single-institution Trial of Carbon-ion Radiotherapy Combined With Granulocyte-macrophage Colony-stimulating Factor for the Treatment of Hepatocellular Carcinoma
Brief Title: Phase II Trial of Carbon-ion Radiotherapy Combined With GM-CSF for the Treatment of Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment was too slow
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Guoliang Jiang, Director the committee of clinical technique, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HCC2016-02
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; carbon-ion radiotherapy; GM-CSF; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carbon-ion radiotherapy with GM-CSF (Experimental): Hypofractionated carbon-ion radiotherapy was prescribed at a dose of 40Gray(Gy) [relative biological effectiveness (RBE)] in 5 fractions for intrahepatic cases away from gastro-intestinal (GI) tract (>1cm) with concurrent GM-CSF 125ug/m2/d, subcutaneous injection d1-28;
  Interventions: Radiation: carbon-ion radiotherapy

INTERVENTIONS:
Radiation: carbon-ion radiotherapy — Hypofractionated carbon-ion radiotherapy was prescribed at a dose of 40Gy RBE in 5 fractions

SUMMARY:
The aim of this research project is to assess the efficacy and toxicity of hypofractionated carbon-ion radiotherapy with concurrent granulocyte-macrophage colony-stimulating factor for the treatment of hepatocellular carcinoma

DETAILED DESCRIPTION:
Golden E.B. et al.in 2015 reported that localized radiotherapy granulocyte-macrophage colony-stimulating factor (GM-CSF) produced objective abscopal responses in solid tumor with metastasises. We hypothesize that hypofractionated carbon-ion radiotherapy combining granulocyte-macrophage colony-stimulating factor (GM-CSF) might improve the clinical response rate and progression-free survival (PFS) in hepatocellular carcinoma. The primary endpoint of the current phase II trial is progression-free survival rate at 2 years, secondary endpoints are overall survival, safety and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed hepatocellular carcinoma (HCC) or clinical diagnosis of HCC according to American association for the study of liver diseases （AASLD）-guidelines or clinical diagnosis criteria based on Alpha Fetoprotein （AFP), and radiological images proposed by Liver Cancer Society, Chinese Anti-Cancer Association;
2. no clinically distant metastasis;
3. the tumor is away from gastro-intestinal (GI) tract (>1cm);
4. Child Push score A,technically unresectable, or medically inoperable; maximal tumor size is less than 10 cm;
5. age ≥ 18 and <80 years of age;
6. Karnofsky Performance Score ≥ 70;
7. No previous invasive cancer (within 5 years before the HCC diagnosis)except for skin non-melanoma cancer or non muscle invasive bladder cancer; Ability to understand character and individual consequences of the clinical trial;
8. Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial;

Exclusion Criteria:

1. Distant metastasis (M1);
2. maximal tumor size is more than 10 cm;
3. tumor invading adjacent gastrointestine (T4);
4. Child push score B or C;
5. Previous hepatic radiotherapy;
6. Severe systemic disorders;
7. Previous malignancy (within 5 years) except for skin non-melanoma cancer or 3-year disease free interval from previous malignancy like in situ cervix cancer or non muscle invasive bladder cancer;
8. Non conformity of the radiotherapy dose distribution when compared to the dose constraints;
9. Psychiatric disorders or any other condition that can make unreliable the informed consent;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of all patients | 2 year
  Time in months measured from treatment initiation until the date of progression or the date of last follow-up.

SECONDARY OUTCOMES:
Overall Survival | 2 year
  Time in months measured from treatment initiation until the date of death or the date of last follow-up.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time interval from the start of carbon-ion radiotherapy to 3 months after the completion of carbon-ion radiotherapy]
Objective responses rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: guo-liang jiang, Dr., Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (2):
- China (2):
  - Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality
  - Shanghai Proton and Heavy Ion Center, Shanghai

IPD SHARING:
Plan to Share IPD: No